CLINICAL TRIAL: NCT07286864
Title: Effects of Outdoor Horseback Riding on Lower Extremity Muscle Strength, Core Stabilization, Balance, Sleep Quality, and Functional Movement Capacity in Healthy Adults
Brief Title: Outdoor Horseback Riding and Its Effects on Muscle Strength, Balance, Sleep, and Movement
Status: Recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Other Study IDs: 25-109
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Sports Physical Therapy; Physical Functional Performance; Horseback Riding
Keywords: Outdoor horseback riding; Sleep quality; Balance; Functional movement; Core stabilization; Lower extremity strength
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Horseback Riders group: Horseback Riders:
  Adults aged 18-65 who have been riding horses outdoors regularly (at least once per week) for a minimum of 6 months. Participants will undergo assessments of lower extremity muscle strength, core stabilization, balance, functional movement, and sleep quality. No experimental interventions are assigned; participants continue their usual riding activities.
- Healthy group (Non-riders / Control Group): Adults aged 18-65 who do not ride horses.Participants will undergo assessments of lower extremity muscle strength, core stabilization, balance, functional movement, and sleep quality.

SUMMARY:
This study aims to investigate the effects of regular outdoor horseback riding on lower extremity muscle strength, core stabilization, balance, functional movement capacity, sleep quality, and overall well-being in healthy adults. Participants with at least 6 months of routine outdoor horseback riding will be compared to non-riders to evaluate differences in physical performance and functional capacity. The study will provide evidence on the potential health benefits of horseback riding.

DETAILED DESCRIPTION:
This observational study will include two groups: a horseback riding group (n=32) and a non-riding control group (n=32). Participants in the riding group must have engaged in outdoor horseback riding at least once per week for a minimum of 6 months. The control group will consist of healthy individuals who do not participate in regular physical activity. At baseline, all participants will undergo the following assessments: Demographic information Lower extremity muscle strength using a digital dynamometer Core stabilization (plank test) Functional movement screening (FMS) Balance assessment (Y-Balance Test Lower Quarter, Modified Functional Reach Test) Sleep quality (Pittsburgh Sleep Quality Index) Overall health-related quality of life (SF-36) Anxiety levels (Beck Anxiety Inventory) All procedures will be performed under standardized conditions with instructions and demonstrations provided to participants. Muscle strength and functional tests will follow established protocols including repetitions, rest intervals, and safety precautions. Balance assessments will be performed barefoot, and reach distances will be normalized for leg length. Data will be analyzed to compare the physical and functional performance, balance, core stabilization, and sleep quality between horseback riders and non-riders. The results will provide insights into the effects of outdoor horseback riding on physical health and functional capacity in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 65 years. Regular outdoor horseback riding for at least 6 months (minimum once per week). Voluntary participation and signed informed consent. Healthy individuals without chronic musculoskeletal, cardiovascular, or neurological diseases.

Cognitive ability to understand instructions and communicate.

Exclusion Criteria:

Any orthopedic, neurological, cardiovascular, or respiratory disease. Diagnosed sleep disorder, anxiety, depression, or other psychiatric conditions. Major surgery within the past 6 months. Pregnancy. Physical or cognitive conditions preventing completion of study protocols. Inability to comply with test procedures or cooperate during assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include healthy adults aged 18-65 years. Participants will be divided into two groups: individuals who have been regularly practicing outdoor horseback riding for at least 6 months (minimum once per week) and individuals who do not participate in horseback riding or regular physical activity. All participants must be able to understand instructions, communicate effectively, and complete the study assessments.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-16 (Estimated)

PRIMARY OUTCOMES:
Lower Extremity Muscle Strength | Single assessment during study visit (1 day)
  Lower extremity muscle strength assessments will be performed using a digital hand-held dynamometer. The force parameters were recorded in kilograms. Isometric muscle strength measurements will be carried out for the following muscle groups: Hip: Flexion, Extension, Abduction, and Adduction Knee: Flexion and Extension Ankle: Plantar flexion, Dorsiflexion For each muscle group, participants will be instructed to maintain maximum isometric muscle contractions that reach equilibrium against the counterforce applied by the researcher, while sustaining the test positions for approximately 3 seconds. Each movement will be performed three times, and the average of these three trials will be considered for evaluation. To minimize fatigue, a rest period of 30-60 seconds will be given between repetitions and 2 minutes between different tests.
Core Stabilization (Assessed using the plank test) | Single assessment during study visit (1 day)
  Participants will be asked to rise by supporting themselves on their elbows and hands, positioned at shoulder level on the mat, while also maintaining support on their toes. During the test, it will be expected that the spine and pelvis remain in a neutral position and that normal breathing is sustained. Participants will be required to maintain this position without descending to the mat, without experiencing pain, and without deviating more than 5 cm in their back, for up to a maximum of 3 minutes. The stopwatch will be started with the command "Start!" and stopped when one of the predetermined termination criteria occurs. The duration will be recorded in seconds, rounded to the nearest whole second.
Functional Movement Screen | Single assessment during study visit (1 day)
  FMS consists of seven test component which are used to evaluate various main movement models.Individuals completed one by one deep squat, high stepping, single line lunge, shoulder mobility, straight leg raises, trunk stability push-ups, rotation stability which are component tests. Subcomponent tests assess asymmetry by measuring the individual bilaterally. Each component test was scored on an ordinal scale (0 to 3 points), with a maximum score of 3, based on the quality of the movement. Less than 3 points indicated that the individual performed some form of compensation or was unable to complete the entire movement.. The scores of the component tests were summed, resulting in a composite score between 0 and 21 points, with a maximum score of 21
Y-Balance Test Score | Single assessment during study visit (1 day)
  YBT, which is performed in the standing position on one leg , is dynamic a test. Participants stood on the footplate in the centre of the Y Balance Test area and then, it was given instruction them that they should maintain a single leg stance while reaching as far as possible with the opposite leg and return to the starting position on the centre platform without losing balance.In the test, individuals were asked to reach the maximum distance in 3 directions (anterior, posteromedial and posterolateral), allowing 3 trials for each leg. The maximum reach distance was recorded for each consecutive trial
Modified Functional Reach Test (MFRT) | Single assessment during study visit (1 day)
  MFRT is a seated version of the original standing test and assesses the limits of balance. The participant sits on a chair with the hips, knees, and ankles flexed at 90 degrees, with the soles of the feet fully in contact with the floor. A horizontal ruler is mounted on the wall at the level of the acromion of the unaffected arm. The starting measurement is taken at the level of the fifth finger when the arm is extended forward at 90 degrees of flexion. The test is performed in three different positions, each consisting of three trials: 1. Reaching forward with the unaffected side facing the wall. 2. Bending to the right with the back against the wall. 3. Bending to the left with the back against the wall. Participants are asked to reach the maximum distance without rotating or touching the wall. After reaching, the position of the fifth finger is marked again, and the distance is measured in centimeters.
Pittsburgh Sleep Quality Index | Single assessment during study visit (1 day)
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions which measures seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
Beck Anxiety Inventory (BAI) | Single assessment during study visit (1 day)
  The Beck Anxiety Inventory (BAI) consists of 21 self-reported items (four-point scale ranging from 0 to 3. p.) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63).
Short Form 36 (SF-36) | Single assessment during study visit (1 day)
  Short Form 36 (SF-36) is a generic self-reported outcome measure that quantifies the quality of life in relation to health status. It is a 36-item valid and reliable evaluation with eight areas covering physical functioning, role limitations brought on by physical issues, bodily pain, general health perceptions, vitality, social functioning, role limitations brought on by emotional issues, and perceived mental health. The SF-36 also contains a single question called "health transition" that measures how respondents feel their over health status has changed over the course of a year. The scores range from 0-100 (the worst possible to the most possible)

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Istinye University, Istanbul
  - Istınye Unıversıtesı, Istanbul
  - İstinye University, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
At this time, there is no finalized plan to share individual participant data (IPD). Data may contain sensitive personal information, and sharing will require additional ethical approvals and anonymization. Decisions regarding data sharing will be made after the study is completed.

REFERENCES:
- [Result] Uldahl M, Christensen JW, Clayton HM. Relationships between the Rider's Pelvic Mobility and Balance on a Gymnastic Ball with Equestrian Skills and Effects on Horse Welfare. Animals (Basel). 2021 Feb 9;11(2):453. doi: 10.3390/ani11020453. PMID 33572205
- [Result] Asgari M, Alizadeh S, Sendt A, Jaitner T. Evaluation of the Functional Movement Screen (FMS) in Identifying Active Females Who are Prone to Injury. A Systematic Review. Sports Med Open. 2021 Nov 22;7(1):85. doi: 10.1186/s40798-021-00380-0. PMID 34807359
- [Result] O'Connor FG, Deuster PA, Davis J, Pappas CG, Knapik JJ. Functional movement screening: predicting injuries in officer candidates. Med Sci Sports Exerc. 2011 Dec;43(12):2224-30. doi: 10.1249/MSS.0b013e318223522d. PMID 21606876
- [Result] Katz-Leurer M, Fisher I, Neeb M, Schwartz I, Carmeli E. Reliability and validity of the modified functional reach test at the sub-acute stage post-stroke. Disabil Rehabil. 2009;31(3):243-8. doi: 10.1080/09638280801927830. PMID 18608433
- [Result] Vazquez Morejon AJ, Vazquez-Morejon Jimenez R, Zanin GB. Beck Anxiety Inventory: psychometric characteristics in a sample from the clinical Spanish population. Span J Psychol. 2014 Oct 28;17:E76. doi: 10.1017/sjp.2014.76. PMID 26055653
- [Result] Demiral Y, Ergor G, Unal B, Semin S, Akvardar Y, Kivircik B, Alptekin K. Normative data and discriminative properties of short form 36 (SF-36) in Turkish urban population. BMC Public Health. 2006 Oct 9;6:247. doi: 10.1186/1471-2458-6-247. PMID 17029646
- [Result] Sipe CL, Ramey KD, Plisky PP, Taylor JD. Y-Balance Test: A Valid and Reliable Assessment in Older Adults. J Aging Phys Act. 2019 Sep 1;27(5):663-669. doi: 10.1123/japa.2018-0330. PMID 30676192
- [Result] Garcia-Pena IM, Gomez AG, Guerrero-Barona E, Moreno-Manso JM, Barrios-Fernandez S. Physical Activity and Sleep Improvements in a Group of Equestrian Therapy Volunteers: A Pilot Study. Evid Based Complement Alternat Med. 2022 Mar 30;2022:5364491. doi: 10.1155/2022/5364491. eCollection 2022. PMID 35399627
- [Result] Thompson Coon J, Boddy K, Stein K, Whear R, Barton J, Depledge MH. Does participating in physical activity in outdoor natural environments have a greater effect on physical and mental wellbeing than physical activity indoors? A systematic review. Environ Sci Technol. 2011 Mar 1;45(5):1761-72. doi: 10.1021/es102947t. Epub 2011 Feb 3. PMID 21291246
- [Result] Peddie L, Gosselin Boucher V, Buckler EJ, Noseworthy M, Haight BL, Pratt S, Injege B, Koehle M, Faulkner G, Puterman E. Acute effects of outdoor versus indoor exercise: a systematic review and meta-analysis. Health Psychol Rev. 2024 Dec;18(4):853-883. doi: 10.1080/17437199.2024.2383758. Epub 2024 Aug 6. PMID 39108077
- [Result] Elmeua Gonzalez M, Sarabon N. Muscle modes of the equestrian rider at walk, rising trot and canter. PLoS One. 2020 Aug 18;15(8):e0237727. doi: 10.1371/journal.pone.0237727. eCollection 2020. PMID 32810165
- [Result] Bystrom A, Egenvall A, Eisersio M, Engell MT, Lykken S, Lundesjo Kvart S. The impact of teaching approach on horse and rider biomechanics during riding lessons. Heliyon. 2025 Jan 14;11(2):e41947. doi: 10.1016/j.heliyon.2025.e41947. eCollection 2025 Jan 30. PMID 39906839
- [Result] Legg K, Cochrane D, Gee E, Macdermid P, Rogers C. Physiological Demands and Muscle Activity of Jockeys in Trial and Race Riding. Animals (Basel). 2022 Sep 8;12(18):2351. doi: 10.3390/ani12182351. PMID 36139208
- [Result] Kim MJ, Kim T, Oh S, Yoon B. Equine Exercise in Younger and Older Adults: Simulated Versus Real Horseback Riding. Percept Mot Skills. 2018 Feb;125(1):93-108. doi: 10.1177/0031512517736463. Epub 2017 Oct 26. PMID 29073822
- [Result] Yu CH, Kim UR, Kwon TK. Fundamental study of basal physical fitness and activities of daily living for the aged in relation to indoor horse riding exercise. Biomed Mater Eng. 2014;24(6):2407-15. doi: 10.3233/BME-141054. PMID 25226941
- [Result] Collado-Mateo D, Lavin-Perez AM, Fuentes Garcia JP, Garcia-Gordillo MA, Villafaina S. Effects of Equine-Assisted Therapies or Horse-Riding Simulators on Chronic Pain: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2020 Aug 31;56(9):444. doi: 10.3390/medicina56090444. PMID 32878327
- [Result] Yu CH, Hong CU, Kang SR, Kwon TK. Analysis of basal physical fitness and lumbar muscle function according to indoor horse riding exercise. Biomed Mater Eng. 2014;24(6):2395-405. doi: 10.3233/BME-141053. PMID 25226940